CLINICAL TRIAL: NCT00427115
Title: Pilot Study of an Exercise an Psycho-Educational Intervention During Allogeneic Stem Cell Transplantation
Brief Title: Multimodal Intervention in Allogeneic Stem Cell Transplantation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: University Hospitals Center for Nursing and Care Research, Copenhagen, Denmark, Copenhagen University Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 01-173/04
Record Dates: First submitted 2007-01-25; First posted 2007-01-26 (Estimated); Last update posted 2008-05-21 (Estimated); Status verified 2008-05

CONDITIONS: Allogeneic Stem Cell Transplantation; Leukemia
Keywords: Patients undergoing allogeneic stem cell transplantations
MeSH Terms: conditions — Leukemia

INTERVENTIONS:
Behavioral: Multimodal exercise and psychosocial program

SUMMARY:
Objective: To evaluate the feasibility and safety of a 4-6 weeks exercise - psycho-educational intervention in patients undergoing allogeneic stem cell transplantation (allo-HCST). The intervention included structured and supervised exercise, relaxation and psycho-educational components. It was hypothesized that the intervention would minimize loss of physical capacity during hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 yrs
* patients undergoing allogeneic stem cell transplantation

Exclusion Criteria:

* recent cardiovascular or pulmonary disease
* abnormal EKG
* psychiatric disorder
* motor function, musculoskeletal or neurological disturbances
* bony metastasis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2005-08; Primary Completion 2007-12 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Physical capacity VO2 max, muscle strength (1RM, Isometric), stair test | Baseline, post

SECONDARY OUTCOMES:
quality of life indices | baseline, post, 3 and 6 months
FACT-An, EORTC, HADS, Mini-Mac, Symptom Assessment form | baseline, post, 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Jarden, MSN PhD stud, Principal Investigator — Copenhagen University Hospital, Denmark; Lis Adamsen, ProfessorPhD, Study Chair — Copehagen University, Faculty of Health Sciences, Denmark
Locations (1):
- Copenhagen University Hospital, Copenhagen, Denmark